CLINICAL TRIAL: NCT00610857
Title: Safety and Efficacy of Combination Biotherapy With High-dose Interferon Alfa-2b and Anti-CTLA4 Monoclonal Antibody for Recurrent Inoperable Stage III or Stage IV Melanoma
Brief Title: Safety and Efficacy of Combination HDI and Anti-CTLA4 for Recurrent Inoperable Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ahmad Tarhini (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Ahmad Tarhini, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 05-125
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anti-CTLA4 monoclonal antibody and HDI (Experimental): Specific Aim #1: Test the hypothesis that the combination of IFNa-2b and anti-CTLA-4 monoclonal antibody will improve the response rate in patients with recurrent inoperable AJCC stage III and stage IV melanoma. Our therapeutic target is achieving, with acceptable toxicity, a 20% or better rate of objective response, CR or PR by RECIST criteria, as compared to the 5% to 10% expected in patients eligible for study. Study size is planned in terms of our primary efficacy endpoint, objective response.
  Interventions: Drug: Anti-CTLA4 monoclonal antibody and HDI

INTERVENTIONS:
Drug: Anti-CTLA4 monoclonal antibody and HDI — One course of therapy consists of three cycles (1 cycle=28days). Anti-CTLA4 monoclonal antibody (15 mg/kg i.v.) will be given during the first cycle only. HDI will be given all three cycles - cycle 1: 20 MU/m2 i.v. on days 0, 1, 2, 3, 4 a week (MTWRF) for 4 weeks; cycle 2: 10 MU/m2 s.c. 3 days a week (MWF) for 4 weeks; and cycle 3: 10 MU/m2 s.c. 3 days a week (MWF) for 4 weeks.
  Response assessment will be carried out at day 56 and day 84. Every patient will receive 3 cycles regardless of response status after the first 2 cycles. However, a patient may be taken off therapy in the event of clinical progression at the discretion of the treating physician.
  Patients without evidence for disease progression after 3 cycles may be offered additional cycles two weeks after completion of the third cycle. Therapy will continue for a maximum of 12 months.
  Other Names: Anti-CTLA4 monoclonal antibody (CP-675,206)

SUMMARY:
To determine the safety and efficacy of the combination of HDI and anti-CTLA-4 monoclonal antibody for patients with recurrent inoperable stage III or stage IV melanoma.

DETAILED DESCRIPTION:
Immunity to melanoma appears to be central to disease control in the adjuvant and advanced disease settings. Spontaneous regression has been reported in melanoma, suggesting a role for host immunity, indirectly supported by the presence of lymphoid infiltrates at primary melanoma associated with tumor regression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a written informed consent obtained prior to the initiation of study procedures.
* Male and female subjects greater than or equal to 18 years of age.
* Patients must have histologically confirmed recurrent stage III or stage IV melanoma (AJCC 6th edition classification). Cutaneous melanoma, ocular or mucosal melanoma will be eligible.
* Patients must have measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST). Baseline measurements must be obtained within 4 weeks prior to initiating therapy.
* Patients must have adequate hematologic, renal, and liver function as evidenced by the following (within 4 weeks prior to starting the study drugs):
* WBC greater than or equal to 3,000/mm3
* Lymphocytes greater than or equal to 1,000/mm3
* Platelets greater than or equal to 100,000/mm3
* Serum Creatinine less than or equal to 1.5 x upper limit of normal (ULN)
* Serum Bilirubin less than or equal to 1.5 x ULN
* Serum AST/ALT less than or equal to 2.5 x ULN
* Serum LDH less than or equal to 2.0 x ULN
* APTT less than < 40 s
* Patients must have fully recovered from any effects of major surgery, and be free of significant detectable infection.
* Patients must not have received any chemotherapy, hormonal therapy, radiotherapy, or biological therapy within the preceding 4 weeks.
* Patients must not have previous therapy with Anti-CTLA4 monoclonal antibodies (including CP-675,206 and MDX-010). Previous therapy with Interferon-alfa 2b in the adjuvant or metastatic setting is allowed. Previous therapy with other biological agents (including vaccines and GM-CSF) is allowed.
* Patients must have ECOG performance status of 0 or 1.
* Patients must not have autoimmune disorders (except vitiligo). Patients with positive titers for autoimmune antibodies are allowed on the study in the absence of history of clinical manifestations of autoimmune disease.
* Patients must not have conditions of immunosuppression or chronic requirement for treatment with systemic steroids, including oral steroids, continuous use of topical steroid creams or ointments, or any inhaled steroid containing inhalers. Patients who discontinue use of these classes of medication for at least 2 weeks are eligible. Treatment with steroids or other immunosuppressant medications is allowed during the study if clinically required to treat side effects related to autoimmunity that may develop secondary to the study agents.
* Patients must be free of brain metastasis by contrast-enhanced CT/MRI scans within 4 weeks prior to starting the study drugs. If known to have prior brain metastases, must not have evidence of active brain disease on two successive MRI evaluations at least 3 months apart (one of which is £ 4 weeks prior to starting the study drugs).
* Female patients of child bearing potential must have a negative pregnancy test, and must not be breast feeding.
* Patients must agree to use effective contraception (both males and females).

Exclusion Criteria

* Serious illnesses, such as: cardiovascular disease (uncontrolled congestive heart failure, hypertension, cardiac ischemia, myocardial infarction, severe cardiac arrhythmia), bleeding disorders, autoimmune diseases, severe obstructive or restrictive pulmonary diseases, active systemic infections, and inflammatory bowel disorders.
* Treatment with mitomycin C or nitrosureas within six weeks prior to study entry.
* Any significant psychiatric disease, medical intervention, or other condition, which in the opinion of the principal investigator, could prevent adequate informed consent or compromise participation in the clinical trial.
* Active infection or antibiotics within one-week prior to study, including unexplained fever (temp > 38.1°C).
* Treatment with anticoagulants, except to keep an indwelling line patent.
* Systemic steroid or other immunosuppressive therapy within 4 weeks of starting the study.
* Treatment with any investigational product within 28 days of registration.
* History of inflammatory bowel disease (e.g. Crohn's disease or ulcerative colitis), celiac disease, or other chronic gastrointestinal conditions associated with diarrhea, or current acute colitis of any origin, or any history of diverticulitis (even a single episode) or evidence of diverticulitis at baseline, including evidence limited to CT-scan only.
* Patients who did not tolerate high-dose interferon-α therapy in the adjuvant setting will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPCI Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Interferon Alfa-2b + Tremelimumab: Patients with stage IV melanoma (cutaneous, uveal, or mucosal) and measurable disease, most who had previously received therapy
Period: Overall Study
Arm/Group | Interferon Alfa-2b + Tremelimumab
Started | 37
Completed | 35
Not Completed | 2
Not completed — Not evaluable for response | 2

BASELINE CHARACTERISTICS:
Population: Patients with stage IV melanoma (cutaneous, uveal, or mucosal) and measurable disease, most who had previously received therapy
Groups:
- Interferon Alfa-2b + Tremelimumab: Patients treated with Tremelimumab 15 mg/kg at start of C1 + IFN-2b IV 20 MU/m2/d for 5 d/wk for 4 weeks; C2 onward- IFN-2b SQ 10MU/m2/d for 3 d/wk for 4 weeks
Arm/Group | Interferon Alfa-2b + Tremelimumab
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 56 [28 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Best Objective Response Rate (BORR)
Description: Intention to treat response rate is estimated by the proportion of patients with a best response of CR, PR, or SD by Response Evaluation Criteria in Solid Tumors [RECIST] version 1.0
Time Frame: Up to 44 months
Population: Patients treated with Tremelimumab 15 mg/kg at start of C1 + IFN-2b IV 20 MU/m2/d for 5 d/wk for 4 weeks; C2 onward- IFN-2b SQ 10MU/m2/d for 3 d/wk for 4 weeks
Measure: Number (90% Confidence Interval); unit: percentage of patients
Groups:
- Interferon Alfa-2b + Tremelimumab: Patients treated withTremelimumab 15 mg/kg at start of C1 + IFN-2b IV 20 MU/m2/d for 5 d/wk for 4 weeks; C2 onward- IFN-2b SQ 10MU/m2/d for 3 d/wk for 4 weeks
Arm/Group | Interferon Alfa-2b + Tremelimumab
Number analyzed (Participants) | 37
percentage of patients | 24 [13 to 36]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from initial treatment date of to date of documented progression of disease progression (TTP)
Time Frame: Up to 44 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Interferon Alfa-2b + Tremelimumab
Number analyzed (Participants) | 37
months | 6.4 [3.3 to 12.1]

3. Secondary Outcome: 1-year Overall Survival (OS)
Description: 1-year survival is the estimated probability of surviving one year expressed as a percent (probability of survival is not probability of dying).
Time Frame: Time from initial treatment date, up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Interferon Alfa-2b + Tremelimumab
Number analyzed (Participants) | 37
percentage of patients | 62 [46 to 78]

4. Secondary Outcome: Median Overall Survival (Point Estimate)
Description: Median overall survival is the (point) estimate of the time corresponding to 50% estimated probability of survival.
Time Frame: Up to 44 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Interferon Alfa-2b + Tremelimumab
Number analyzed (Participants) | 37
months | 21 [9.5 to NA] — Upper bound of the CI was not reached

ADVERSE EVENTS:
Time Frame: 5 years.
Description: Includes adverse events that were considered either study treatment-related or unrelated.
Groups:
- Interferon Alfa-2b + Tremelimumab (Related and Unrelated AEs): Patients treated withTremelimumab 15 mg/kg at start of C1 + IFN-2b IV 20 MU/m2/d for 5 d/wk for 4 weeks; C2 onward- IFN-2b SQ 10MU/m2/d for 3 d/wk for 4 weeks per cycle.
Arm/Group | Interferon Alfa-2b + Tremelimumab (Related and Unrelated AEs)
Serious Adverse Events (participants affected / at risk) | 15/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Alfa-2b + Tremelimumab (Related and Unrelated AEs) (N=37)
Pain, Abdomen NOS (Blood and lymphatic system disorders) | 1
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Cardiac disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (General disorders) | 1
Vomiting (Skin and subcutaneous tissue disorders) | 1
Renal failure (Endocrine disorders) | 1
Fatigue (asthenia, lethargy, malaise) (Gastrointestinal disorders) | 1
Ulceration (Gastrointestinal disorders) | 1
Thrombosis/thrombus/embolism (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Hemorrhage, CNS (Blood and lymphatic system disorders) | 1
Supraventricular and nodal arrhythmia, Atrial fibrillation (Metabolism and nutrition disorders) | 1
Diarrhea (Nervous system disorders) | 1
Bronchospasm, wheezing (General disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Renal and urinary disorders) | 1
Secondary Malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
GGT (gamma-Glutamyl transpeptidase) (Vascular disorders) | 1
Encephalopathy (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Alfa-2b + Tremelimumab (Related and Unrelated AEs) (N=37)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 4
Hemoglobin (Blood and lymphatic system disorders) | 10
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 13
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 19
Hypertension (Cardiac disorders) | 3
Sweating (diaphoresis) (General disorders) | 6
Insomnia (General disorders) | 9
Weight loss (General disorders) | 11
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 27
Rigors/chills (General disorders) | 29
Fatigue (asthenia, lethargy, malaise) (General disorders) | 36
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 6
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 6
Pruritus/itching (Skin and subcutaneous tissue disorders) | 23
Rash/desquamation (Skin and subcutaneous tissue disorders) | 26
Dehydration (Gastrointestinal disorders) | 3
Gastrointestinal (Gastrointestinal disorders) | 3
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 13
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 17
Diarrhea (Gastrointestinal disorders) | 21
Anorexia (Gastrointestinal disorders) | 25
Nausea (Gastrointestinal disorders) | 29
Infection with normal ANC or Grade 1 or 2 neutrophils, Upper airway NOS (Infections and infestations) | 4
Edema: limb (Blood and lymphatic system disorders) | 5
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 6
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 8
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 9
Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 4
Mood alteration, Agitation (Nervous system disorders) | 3
Neuropathy: motor (Nervous system disorders) | 4
Neuropathy: sensory (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 6
Mood alteration, Depression (Nervous system disorders) | 7
Neurology (Nervous system disorders) | 8
Mood alteration, Anxiety (Nervous system disorders) | 12
Pain, Extremity-limb (General disorders) | 6
Pain - Other (General disorders) | 7
Pain, Back (General disorders) | 8
Pain, Abdomen NOS (General disorders) | 10
Pain, Head/headache (General disorders) | 12
Pain, Muscle (General disorders) | 16
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes